CLINICAL TRIAL: NCT04480320
Title: Sonography-guided Pericapsular Nerve Group Block for Hip Arthroplasty
Brief Title: Sonography-guided Pericapsular Never Group Block for Hip Arthroplasty
Acronym: QUASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, MD, PhD, Vice-Director in Dept Anesth & Pain, Professor, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-2020-085-01
Record Dates: First submitted 2020-07-02; First posted 2020-07-21 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Arthroplasty; Nerve Block; Analgesia
Keywords: Pericapsular Nerve Group; PENG; hip arthroplasty; Postoperative analgesia; quadriceps strength
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nerve group block (Experimental)
  Interventions: Procedure: pericapsular nerve group block
- Saline placebo group (Placebo Comparator)
  Interventions: Procedure: pericapsular nerve group block

INTERVENTIONS:
Procedure: pericapsular nerve group block — Branches of both the FN and ON provide innervation to the anterior hip capsule. High and low branches of FN provided the majority of innervation to the lateral and superomedial hip capsule. The AON innervates the medial capsule.Both of the nerve close to the periosteum between the iliopubic eminence and AIIS ,by using ultrasound guided technique,these sites can be potential bony landmarks provid approch to the nerve group.

SUMMARY:
In this study, the investigator will examine the efficacy of Pericapsular nerve group (PENG) block in hip arthroplasty as a post-operative pain management technique, study the analgesia, opioid-sparing effects and motor-blocking effects of the PENG block

DETAILED DESCRIPTION:
PENG Block group (PG) will receive 0.5%Ropivacaine in 20 ml of saline. Sham Block group (SG) will receive 20 ml of saline Patient will be sedated with IV midazolam before nerve block. After peripheral nerve block ,general anesthesia will be conducted using sufentanyl, propofol and rocuronium for induction and propofol and sevoflurane for maintenance. Tests will be operated after procedure，and recorded up to 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip arthroplasty

Exclusion Criteria:

* allergy to local anesthetics
* infection at the injection site
* patients receiving opioids for chronic analgesic therapy
* other lower limb neuropathies
* inability to comprehend visual analog scale (VAS)
* preexist cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Highest VAS score in recovery room | before recovery room discharge(up to 2 hours after surgery end)
  Highest VAS score reported in recovery room,patient will be asked questions to measure the highest VAS score experienced in the recovery room before discharge. If the patient had a unexpected long stay at recovery room, the question will be asked at the time point "2 hours after surgery end"

SECONDARY OUTCOMES:
VAS at rest | day0 ,day1 ,day2
  VAS pain score while patient at rest
highest VAS at period | day0 ,day1 ,day2
  highest VAS reported at follow up period
quadriceps strength | day0 , day1 ,day2
  Measure quadriceps strength peak value at different time point
total opioid consumption | up to 2 days after surgery
PONV rate | day0 ,day1 ,day2
  postoperative nausea and vomit
Fall incident happened | up to 2 days after surgery
  Record the fall incident happened,fall is defined as patinent accidently fall to the ground.
Nerve block range | day0 , before discharge from PACU(up to 2 hours after surgery end)
  A cotton yarn with ethanol will be put on both the surgical and nonsurgical leg to evaluate the cold sensation lost after nerve block.Skin sensation lost will be tested at lateral thigh,medial thigh,front thigh and lateral claf

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng J, Pan D, Zheng B, Ruan X. Preoperative pericapsular nerve group (PENG) block for total hip arthroplasty: a randomized, placebo-controlled trial. Reg Anesth Pain Med. 2022 Mar;47(3):155-160. doi: 10.1136/rapm-2021-103228. Epub 2021 Dec 6. PMID 34873023